CLINICAL TRIAL: NCT06216288
Title: The Effects of Combined Lumbar Traction and Repeated Back Extension Exercise on H-Reflex, Pain, and Disability in Patients With Lumbosacral Radiculopathy
Brief Title: Effect of Combined Lumbar Traction and Repetitive Back Extension Exercise on H-reflex in Lumbosacral Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-reflex in Radiculopathy
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lumbosacral Radiculopathy; McKenzie Derangement Syndrome
Keywords: H-reflex; radiculopathy; McKenzie; Lumbar traction
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: participants will be assigned to one of the 2 groups: either the control group receiving McKenzie repeated back extension exercise or the experimental group receiving combined McKenzie and Lumbar traction
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repeated back extension exercise (McKenzie) (Active Comparator): Repeated back extension exercise as described by McKenzie in prone position was performed of three sets of ten repetitions with one minute rest between the sets. The patient was asked to reach the maximum extension possible in all attempts and maintain this position for one second. The intervention was done 3 times per week for 6 weeks.
  Interventions: Other: Repeated back extension exercise (McKenzie)
- Combined mechanical lumbar traction and repeated back extension exercise (McKenzie) (Experimental): Participants allocated to mechanical lumbar traction received the McKenzie approach described above in combination with mechanical lumbar traction. The traction was applied using a 3D ActiveTrac table which is a motorized split table. Participants were placed in prone position and static traction was applied for 15 minutes at an intensity of 40% to 60% of the participant's body weight. At the end of traction intervention, participants continued with the McKenzie repeated back extension exercise intervention. The intervention was done 3 times per week for 6 weeks.
  Interventions: Other: Repeated back extension exercise (McKenzie); Device: Mechanical traction

INTERVENTIONS:
Other: Repeated back extension exercise (McKenzie) — repetitive back extension exercises in prone position with 1 minute hold on maximal back extension. 3 sets of 10 repetitions with 1 minute break between sets. The intervention was done 3 times per week for 6 weeks.
  Other Names: McKenzie Back Extension Approach
Device: Mechanical traction — The traction was applied using a 3D ActiveTrac table. This motorized split table applied static traction to the lumbar spine with the participant in a prone position. The intensity of the force of traction was 40% to 60% of the participant's body weight applied for 15 minutes. The intervention was done 3 times per week for 6 weeks.
  Other Names: mechanical lumbar traction
  Arms: Combined mechanical lumbar traction and repeated back extension exercise (McKenzie)

SUMMARY:
The aim of the study is to investigate the effect of performing combined lumbar traction and repeated back extension exercise (McKenzie) on soleus H-reflex, pain, and disability in patients with lumbosacral radiculopathy. The main question that it aims to answer is:

Does the combination of lumbar traction and back extension exercise (McKenzie) improves soleus H-reflex, pain, and function in patient with lumbosacral radiculopathy? participants will be randomized into 2 groups: one group will include repeated back extension exercise (McKenzie Approach) without mechanical traction and the other group will include the same but in combination with mechanical traction.

DETAILED DESCRIPTION:
Repeated back extension exercises as described by McKenzie from prone position has been widely suggested for patients with lumbosacral radiculopathy (LSR). It has been reported to decrease radicular symptoms which could be due to the decompression effect of this exercise on the compromised nerve root. Moreover, mechanical traction have a debatable effect on lumbosacral patients with little evidence that supports its effectiveness. Thus, the investigators hypothesize that performing a combination of lumbar traction and repeated back extension exercise will improve the soleus H-reflex, pain, and function of lumbosacral radiculopathy patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with chronic unilateral lumbosacral radiculopathy (more than 3 months duration)
2. Age:35- 60 years
3. Both male and female
4. People with L5-S1 postero-lateral disc herniation or protrusion.
5. people with positive straight leg raise

Exclusion Criteria:

1. Subjects with lumbosacral Surgery.
2. Subjects with stenosis or scoliosis.
3. Subjects with cardiac problem or cancer.
4. Subjects with peripheral neuropathy.
5. Subjects with upper motor neuron injury.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Soleus H-reflex amplitude | At baseline and 6 weeks
  amplitude in millivolts (mV)
Soleus H-reflex latency | At baseline and 6 weeks
  latency in milliseconds (ms)

SECONDARY OUTCOMES:
Numerical Pain Intensity Scale | At baseline and 6 weeks
  in numbers, the score ranges from 0 to10.
Oswestry Disability Index (ODI) | At baseline and 6 weeks
  in numbers, the score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Melhat, PhD, Study Director — Cairo University
Locations (1):
- Ahmed ElMelhat [aelmelhat], Cairo, Egypt

REFERENCES:
- [Background] Al-Abdulwahab S. Back extension exercises decompress the spinal root and improve standing mobility in patients with sub-acute lumbosacral radiculopathy. Somatosens Mot Res. 2016 Sep-Dec;33(3-4):196-199. doi: 10.1080/08990220.2016.1251895. Epub 2016 Nov 13. PMID 27838950
- [Background] Vanti C, Saccardo K, Panizzolo A, Turone L, Guccione AA, Pillastrini P. The effects of the addition of mechanical traction to physical therapy on low back pain? A systematic review with meta-analysis. Acta Orthop Traumatol Turc. 2023 Jan;57(1):3-16. doi: 10.5152/j.aott.2023.21323. PMID 36939359
- [Background] Thackeray A, Fritz JM, Childs JD, Brennan GP. The Effectiveness of Mechanical Traction Among Subgroups of Patients With Low Back Pain and Leg Pain: A Randomized Trial. J Orthop Sports Phys Ther. 2016 Mar;46(3):144-54. doi: 10.2519/jospt.2016.6238. Epub 2016 Jan 26. PMID 26813755